CLINICAL TRIAL: NCT01228812
Title: An Observational Study of Physical Activity Behavior of Swiss Rheumatoid Arthritis Patients and Healthy Matched Controls
Brief Title: Physical Activity Behavior of Rheumatoid Arthritis Patients and Healthy Controls
Status: Completed | Type: Observational
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Yves Henchoz, Principal Investigator, Research Officer, University of Lausanne
Other Study IDs: PR_AP
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis, physical activity
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RA patients: Patients with Rheumatoid Arthritis
- Healthy subjects: Healthy subjects matched for age and sex

SUMMARY:
The purpose of the study is to compare physical activity behaviour of rheumatoid arthritis patients with healthy matched controls.

ELIGIBILITY:
Inclusion Criteria (RA patients):

* Rheumatoid arthritis
* Functional classes I, II and III
* Age 40 to 80 years
* Stable disease activity
* Stable DMARDS last 3 months

Exclusion Criteria (RA patients):

* Functional classes IV
* Inflammatory flare

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients from the RA patients group will be selected in the Rheumatology Department of the Centre Hospitalier universitaire Vaudois in Lausanne. Healthy matched controls will be randomly selected from a cohort study conducted in Lausanne.
Sampling Method: Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Physical activity | Up to 4 weeks
  PAFQ

SECONDARY OUTCOMES:
Functional status | Up to 4 weeks
  HAQ
Pain | Up to 4 weeks
  VAS
Fatigue | Up to 4 weeks
  VAS
Disease activity | Up to 4 weeks
  DAS 28

CONTACTS AND LOCATIONS:
Overall Officials: Alexander KL So, PhD, FRCP, Study Director — Université de Lausanne, Service de Rhumatologie, Département de l'Appareil Locomoteur, Lausanne, Suisse; Yves Henchoz, PhD, Principal Investigator — Université de Lausanne, Service de Rhumatologie, Département de l'Appareil Locomoteur, Lausanne, Suisse; Jean Dudler, PD, MER, Study Chair — Université de Lausanne, Service de Rhumatologie, Département de l'Appareil Locomoteur, Lausanne, Suisse; François Bastardot, MD, Study Chair — Etude CoLaus, Centre Hospitalier Universitaire Vaudois, Lausanne; Peter Vollenweider, MD, Study Chair — Etude CoLaus, Centre Hospitalier Universitaire Vaudois, Lausanne; Idris Guessous, MD, Study Chair — Unité d'Epidémiologie Populationnelle, Département de médecine communautaire et de premier recours, Hôpitaux Universitaires de Genève
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Département de l'Appareil Locomoteur, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henchoz Y, Bastardot F, Guessous I, Theler JM, Dudler J, Vollenweider P, So A. Physical activity and energy expenditure in rheumatoid arthritis patients and matched controls. Rheumatology (Oxford). 2012 Aug;51(8):1500-7. doi: 10.1093/rheumatology/kes067. Epub 2012 Apr 25. PMID 22539478